CLINICAL TRIAL: NCT07275229
Title: Efficacy and Safety of Irregular Pulsed Radiofrequency (Sluijter-Teixera Poisson) Versus Regular Pulsed Radiofrequency to the Gasserian Ganglion for Treatment of Primary Trigeminal Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mamdouh Ahmed, Assistant lecture, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: soh-Med-25-11-4MD
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Trigeminal Neuralgia
Keywords: radiofreqency for treatment of trigeminal neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irregular pulsed radiofrequency STP group (Experimental)
  Interventions: Procedure: Irregular pulsed Radiofrequency
- Regular pulsed radiofrequency group (Active Comparator)
  Interventions: Procedure: Regular pulsed Radiofrequency

INTERVENTIONS:
Procedure: Irregular pulsed Radiofrequency — irregular pulsed radiofrequency applied to gasserian ganglion for primary trigeminal neuralgia
  Arms: Irregular pulsed radiofrequency STP group
Procedure: Regular pulsed Radiofrequency — Regular pulsed radiofrequency applied to gasserian ganglion for primary trigeminal neuralgia
  Arms: Regular pulsed radiofrequency group

SUMMARY:
This study aims to compare between the Efficacy and safety of irregular pulsed radiofrequency STP versus regular pulsed radiofrequency to the gasserian ganglion for treatment of primary trigeminal neuralgia.

DETAILED DESCRIPTION:
Trigeminal neuralgia is a severe pain condition characterized by transient, paroxysmal, electric shock-like pain occurring in areas supplied by the trigeminal nerve. The incidence of trigeminal neuralgia increases with advancing age and has a substantial negative impact on quality of life, often leading to psychological distress.

Pharmacological therapy represents the primary treatment modality for most patients with trigeminal neuralgia. Surgical and interventional procedures, including microvascular decompression, partial sensory rhizotomy, radiofrequency therapy, glycerol rhizolysis, balloon compression, and gamma knife surgery, are generally reserved for patients who are resistant or intolerant to medical treatment. Each of these modalities has specific advantages and limitations, and no single ideal surgical treatment has been established.

Pulsed radiofrequency (PRF) is considered one of the least destructive neuromodulation techniques. It stimulates the gasserian ganglion using pulsed electrical current while maintaining tissue temperature below 42°C. The pulsed current is delivered intermittently, allowing heat dissipation and minimizing neural tissue damage. Patients who respond favorably to PRF often experience significant improvement in pain and quality of life; however, conventional PRF has been associated with limited efficacy and a shorter duration of pain relief compared to continuous radiofrequency techniques.

Several modifications have been introduced to enhance PRF effectiveness, including adjustments in output voltage and pulse delivery parameters. Despite these modifications, achieving an optimal balance between efficacy and safety remains challenging.

The Slijter-Teixeira Poisson (STP) mode of pulsed radiofrequency utilizes a Poisson distribution pattern for energy delivery, allowing pulses to be more evenly and precisely distributed. This approach aims to optimize therapeutic outcomes while minimizing heat generation and tissue injury. The STP mode provides shorter pulse widths and a higher coefficient of variance, which may enhance treatment effectiveness without increasing neurodestructive effects.

Accordingly, this study is designed to compare the efficacy and safety of regular pulsed radiofrequency and STP-mode pulsed radiofrequency applied to the gasserian ganglion in patients with primary trigeminal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary trigeminal neuralgia according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)
* Age between 18 and 75 years
* Severe trigeminal neuralgia not adequately relieved by conservative medical therapy, including carbamazepine or oxcarbazepine
* Numeric Rating Scale (NRS-11) pain score of 7 or higher prior to the procedure
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Secondary trigeminal neuralgia, including trigeminal neuralgia attributed to space-occupying lesions or multiple sclerosis
* Infection at the puncture site
* History of psychiatric disease
* Clinically significant abnormalities in routine laboratory tests, including hepatic, renal, or coagulation function, or abnormalities on electrocardiogram or chest X-ray
* Serious systemic diseases, including uncontrolled hypertension or diabetes mellitus, or cardiac dysfunction classified as New York Heart Association class II-III
* History of narcotic substance abuse
* Previous treatment with continuous radiofrequency to the gasserian ganglion or peripheral branches, glycerol rhizolysis, balloon compression, gamma knife surgery, or other neuroablative procedures
* Previous microvascular decompression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | day 1 after 1 and 2 weeks, and after 1, 2, 3 and 6 months following the procedure
  • Pain intensity of the attacks using VAS (''0'' no pain to ''10'' worst possible pain) day 1, after 1and 2 weeks and after 1,2,3 and 6 months. And dose of carbamazepine or oxcarbazepine will be recorded on day 1 after 1 and 2 weeks, and after 1, 2, 3 and 6 months following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Mohamed, assistant professor, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided